CLINICAL TRIAL: NCT04445311
Title: Use of Ivermectin as a Therapeutic Option for Patients With COVID-19
Brief Title: Ivermectin in Treatment of COVID-19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Waheed Shouman, professor of chest diseases, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZU-IRB#6151/31-5-2020
Record Dates: First submitted 2020-06-19; First posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: COVID
MeSH Terms: interventions — Ivermectin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivermectin group (Experimental): group that will receive ivermectin plus standard of care ttt
  Interventions: Drug: Ivermectin
- Control group (No Intervention): group that will receive standard of care ttt

INTERVENTIONS:
Drug: Ivermectin — 3 successive days ttt of ivermectin started within 48 hours of symptoms
  Arms: Ivermectin group

SUMMARY:
confirmed cases with COVID-19 will receive ivermectin as a therapeutic option as well as standard of care treatment and will be compared to those that will receive only standard of care ttt

ELIGIBILITY:
Inclusion Criteria:

COVID-19 patients during period of the study more than 18 years old

Exclusion Criteria:

refuse to participate pregnancy or lactation hypersensitivity to ivermectin receive any drug with interaction with ivermectin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05-31 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-08-15 (Estimated)

PRIMARY OUTCOMES:
time to be symptoms free | within 21 days after enrollment
  duration from day 1 symptoms till 3 days without symptoms

SECONDARY OUTCOMES:
hospitalization | within 21 days after enrollement
  need hospital admission
Mechanical ventilation | within 21 days after enrollement
  need mechanical ventilation
length of stay | within one month days after enrollement
  days spent in hospital
mortality | within one month days after enrollement
  survived or died

CONTACTS AND LOCATIONS:
Locations (1):
- Waheed Shouman, Zagazig, Sharqia Province, Egypt